CLINICAL TRIAL: NCT01926964
Title: Impact of Recurrence Score® on Recommendations for Adjuvant Treatment in Patients With ER-positive Breast Cancer
Brief Title: Adjuvant Treatment Recommendation and Oncotype DX® in Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: SAKK 26/10; 01-086 (Other: Genomic Health Inc.)
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: Adjuvant treatment recommendation; Early breast cancer; Oncotype DX; Genetic profiling
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Early breast cancer patients: Patients with ER-positive, HER2 negative, pN0 or pN1a and resected primary breast cancer R0 resection.

SUMMARY:
Oncotype DX® is likely to become more widely used in Europe as well as in Switzerland. The test is currently not reimbursed by the Swiss health insurances.

The proposed study will investigate to what extent adjuvant treatment recommendations in breast cancer patients with an ER-positive tumor, made by Swiss tumor boards, are based on conventional factors, and whether the recommendations would change, when RS results from the Oncotype DX® test were available.

In addition this study approaches the dilemma of adding adjuvant CT to adjuvant endocrine therapy in a systematic fashion. In this study, the St. Gallen consensus 2009 (with a minor update from the 2011 consensus, is used to predefine the patients suitable for endocrine therapy or chemo-endocrine therapy. Once results of this study are available they may help to better integrate Oncotype DX® with other factors. Currently, it is unclear how the different factors should be integrated into one recommendation.

This study will provide data on the usefulness of this test for the two patient groups which are suitable for hormone therapy only and for those who are considered for hormone plus chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

- Patients screening criteria

1. ≥ 18 years old female patients.
2. Resected primary breast cancer (R0 resection).
3. ER-positive breast cancer (defined as at least 10% ER-positive malignant cells).
4. HER2 negativity by IHC (0 or 1+) or by FISH (negative if ratio is ≤ 2.0).
5. pN0 or pN1a (1-3 positive nodes) by sentinel procedure or axillary dissection.

All patients matching the screening criteria should be recorded consecutively in the patient screening and enrollment list.

Patients inclusion criteria for baseline data collection

1. Signed informed consent form for participation to the baseline data collection.

   In addition, the following information must be available from the pathology report:
2. Estimation of the pathologic maximum tumor diameter (in mm).
3. Results of ER positive tumor cells (in %) and of PgR positive tumor cells (in %) of the invasive component.
4. Proliferation rate by Ki-67 staining (MIB-1 antibody) in %.
5. Result of modified Bloom-Richardson-Elston (BRE) Grading (Grade 1, 2 or 3).

Patients eligibility criteria for participation to the study Inclusion criteria

1. Signed informed consent form for participation to the study SAKK 26/10.
2. The patient is considered suitable to receive adjuvant chemotherapy (ie no medical contraindications to chemotherapy).
3. Invasive breast cancer tissue is available to prepare 39 sections (35 unstained + 4 H&E stained slides, thickness of 5 µm).
4. Performance Status: 0 or 1.

Exclusion criteria

1. Pregnancy
2. Bilateral invasive breast cancer
3. cT4 and pT4 tumors.
4. Patient with a current psychiatric or medical diagnosis that would interfere with her ability to participate in this study.
5. Known metastatic breast cancer (M1).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ER-positive, HER2 negative, pN0 or pN1a and resected primary breast cancer R0 resection.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The decision change between the first and second tumor board adjuvant treatment recommendation | 1 month

SECONDARY OUTCOMES:
The decision change between first and second shared decision about adjuvant treatment | 3 weeks
The decision change between first shared decision and treatment actually given | Between 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Pestalozzi, Prof, Study Chair — University Hospital, Zürich; Stefan Aebi, Prof., Study Chair — Luzerner Kantonsspital
Locations (19):
- Switzerland (19):
  - Kantonsspital Baden, Baden
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Klinik Engeried / Praxis Oncocare, Bern
  - Inselspital, Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Frauenfeld / Brustzentrum Thurgau, Frauenfeld
  - Kantonsspital Freiburg, Fribourg
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital Olten, Olten
  - Tumorzentrum ZeTUP, Sankt Gallen
  - Kantonsspital St. Gallen, Sankt Gallen
  - SpitalSTS AG Simmental-Thun-Saanenland, Thun
  - Kantonsspital Winterthur, Winterthur
  - Brust-Zentrum Seefeld, Zurich
  - Triemli Stadtspital / Frauenklinik, Zurich
  - UniversitaetsSpital, Zurich

REFERENCES:
- [Result] Pestalozzi BC, Tausch C, Dedes KJ, Rochlitz C, Zimmermann S, von Moos R, Winterhalder R, Ruhstaller T, Mueller A, Buser K, Borner M, Novak U, Nussbaum CU, Seifert B, Bigler M, Bize V, Vilei SB, Rageth C, Aebi S; Swiss Group for Clinical Cancer Research (SAKK). Adjuvant treatment recommendations for patients with ER-positive/HER2-negative early breast cancer by Swiss tumor boards using the 21-gene recurrence score (SAKK 26/10). BMC Cancer. 2017 Apr 13;17(1):265. doi: 10.1186/s12885-017-3261-1. PMID 28407750